CLINICAL TRIAL: NCT06198764
Title: A Multicenter, Randomized, Open, Parallel Controlled Clinical Study to Evaluate the Efficacy and Safety of Colistimethate Sodium for Injection in the Treatment of Carbapenem Resistant Gram-negative Infections in Chinese Adults.
Brief Title: A Clinical Trial for the Treatment of Carbapenem Resistant Gram-negative Bacterial Infection With Colistimethate Sodium for Injection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQD3519-CS-01
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — colistinmethanesulfonic acid; Injections; Meropenem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colistimethate sodium for Injection + Meropenem (Experimental): Intravenous infusion of colistimethate sodium for injection for 7-14 days. Meropenem intravenous infusion once every 8 hours or 12 hours.
  Interventions: Drug: Colistimethate sodium for injection; Drug: Meropenem for Injection
- Coly-Mycin® M Parenteral + Meropenem (Active Comparator): Intravenous infusion of Coly-Mycin® M Parenteral for 7-14 days. Meropenem intravenous infusion once every 8 hours or 12 hours.
  Interventions: Drug: Meropenem for Injection; Drug: Coly Mycin M Injectable Product

INTERVENTIONS:
Drug: Colistimethate sodium for injection — Colistimethate Sodium for Injection is the Prodrug of Polymyxin E, which is hydrolyzed into Polymyxin E after entering the human body to play a bactericidal role.Polymyxin selectively acts on gram-negative aerobic bacteria with hydrophobic outer membrane, leading to cell death by destroying the cell membrane.
  Arms: Colistimethate sodium for Injection + Meropenem
Drug: Meropenem for Injection — Meropenem is a broad-spectrum carbapenem antibiotic that inhibits the synthesis of bacterial cell walls by penetrating the cell wall and reaching its target, the penicillin-binding protein, to ultimately produce antibacterial effects.
Drug: Coly Mycin M Injectable Product — Coly Mycin M is the originally marketed colistimethate sodium for injection.
  Arms: Coly-Mycin® M Parenteral + Meropenem

SUMMARY:
A clinical study to evaluate Colistimethate Sodium for Injection combination with Meropenem versus Coly-Mycin® M Parenteral combined with Meropenem in the treatment of Carbapenem resistant gram-negative bacteria infection. A total of 80 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old (based on the signing time of the informed consent form).
* The subject (or their guardian) voluntarily signs an informed consent form.
* Clinical diagnosis confirmed carbapenem resistant Gram negative bacterial infections, including hospital-acquired bacterial pneumonia (HAP) / ventilator-associated bacterial pneumonia (VAP), complicated urinary tract infection (cUTI) , complicated intra-abdominal infection (cIAI), and bloodstream infection (BSI) subjects (minimum disease criteria refer to each additional inclusion criteria)
* Cultivate a Gram negative bacterium identified as carbapenem resistant within 5 days before or during the screening period (mainly including carbapenem resistant Enterobacteriaceae, carbapenem resistant Acinetobacter baumannii, and carbapenem resistant Pseudomonas aeruginosa), and the Gram negative bacteria showed drug resistance to carbapenems in vitro drug sensitive test. In this study, gram-negative bacteria resistant to carbapenems also included strains with bacterial drug sensitivity displayed as "intermediate", that is, resistant bacteria include strains that are intermediate and resistant to carbapenem antibiotics.
* Within 72 hours before randomization, for those who have previously received empirical antimicrobial treatment, the duration of antimicrobial treatment (excluding polymyxin antibiotics) does not exceed 24 hours or the treatment exceed 48 hours but the infection symptoms/signs still exist or become worsen.
* HAP/VAP subjects are required to meet:

  1. Patients with acute pulmonary parenchymal infection who have been hospitalized for more than 48 hours or discharged for less than 7 days, or have received mechanical ventilation through oral or nasal tracheal intubation for at least 48 hours;
  2. Chest X-ray examination (or computed tomography) obtained within 72 hours before randomization shows new infiltrating lesions or progression of existing lesions;
  3. Individuals with at least 2 of the following clinical symptoms/signs:

     1. New occurrence cough；
     2. Produce purulent sputum or tracheal secretions；
     3. The auscultation results are accord with pneumonia/lung consolidation (such as wet rale, dry rale, bronchial breath sound, egophony, dull percussion note);
     4. Difficulty in breathing, shortness of breath (respiratory rate>25 breaths/minute), or hypoxemia (oxygen saturation< 90% when breathing indoor air at standard atmospheric pressure or arterial blood oxygen partial pressure (PaO2) obtained through arterial blood gas (ABG)<60 mmHg);
     5. The oxygenation index (arterial partial pressure of oxygen/percentage of inhaled oxygen concentration (PaO2/FiO2)) deteriorates, requiring urgent changes in ventilator support status or changes in positive end expiratory pressure ventilation volume.
  4. Within 72 hours before the first dose of study drug, the subject is required to take appropriate respiratory specimens (such as sputum, respiratory secretions, culture samples, etc.)
  5. With at least one of the following evidence of systemic inflammatory reactions:

     1. Recorded fever (oral temperature ≥ 38 ℃ or axillary temperature ≥ 37.5 ℃) or hypothermia (rectal/core temperature ≤ 35 °C);
     2. Peripheral blood leukocyte count ≥ 10000/mm ^3 or peripheral blood leukocyte count ≤ 4500/mm ^3 or peripheral blood rod-shaped granulocytes >15%.
* CUTI subjects with/without pyelonephritis are required to meet:

  1. Urinary routine examination shows pyuria, i.e. non centrifuge urine examination ≥ 10 WBC/µ l, centrifuge urine examination white blood cell count (WBC) >5/HPF, or urine routine WBC higher than the upper limit of normal values of each participating unit;
  2. Individuals with at least 2 of the following clinical symptoms or signs:

     1. Fever with or without chills or chills. Acute pyelonephritis must have signs of fever.
     2. Lateral abdominal pain or pelvic pain;
     3. Nausea or vomiting;
     4. Difficulty of urinating, frequent urination, urgency or pain in urination;
     5. There is tenderness or percussion pain in the costovertebral angle during physical examination.
  3. The subject must have at least one of the following basic diseases or conditions with abnormal urinary tract structure or function(excluding acute pyelonephritis):

     1. Urinary tract obstruction (renal stones, renal fibrosis);
     2. Functional/anatomical abnormalities of the genitourinary tract (including anatomical abnormalities or neurogenic bladder) or residual urine volume after urination ≥ 100 mL;
     3. Urinary retention, including those caused by benign prostatic hypertrophy;
     4. Patients with renal diseases such as glomerulonephritis and nephrotic syndrome;
     5. It is known that patients meet the requirements of 30 mg/g<urinary microalbumin/creatinine ratio ≤ 300 mg/g with diabetes nephropathy.
  4. Within 72 hours before the first dose of study drug, subjects are required to take clean mid section urine, with a bacterial colony count in urine culture greater than 105 CFU/mL.
* CIAI subjects are required to meet:

  1. Subjects must arrange or have completed open surgery, laparoscopic surgery, or percutaneous drainage of abdominal abscesses for the diagnosis and treatment of cIAI within 24 hours of enrollment or within 24 hours of administering the first dose of antibiotics;
  2. For subjects enrolled before surgery, study medication can only be administered when there is a high suspicion or diagnosis of intra-abdominal infection, and baseline intra-abdominal culture specimens from the infected site are planned to be obtained;
  3. Appearance of one or more systemic symptoms or signs of cIAI, such as fever, hypotension, abdominal pain, nausea and vomiting, abdominal lumps found during physical examination, and changes in mental state.
  4. With at least one of the following evidence of systemic inflammatory response:

     1. Recorded fever (oral temperature ≥ 38 ℃ or axillary temperature ≥ 37.5 ℃) or hypothermia (rectal/core temperature ≤ 35 °C);
     2. Peripheral blood leukocyte count ≥ 10000 /mm^3 or peripheral blood leukocyte count ≤ 4500 /mm^3 or peripheral blood rod-shaped granulocytes >15%.
* BSI subjects are required to meet:

  1. At least one of blood culture tests conducted was positive within 5 days prior to screening, indicating the presence of Gram negative bacteria. This research can include participants with multiple microbial(Including carbapenem resistant Gram negative bacteria) infections. (Note: This study plans to include patients with primary BSI, defined as pathogenic microorganisms with positive blood culture that are not associated with other infection sites.)
  2. With at least one of the following evidence of systemic inflammatory response:

     1. Recorded fever (oral temperature ≥ 38 ℃ or axillary temperature ≥ 37.5 ℃) or hypothermia (rectal/core temperature ≤ 35 °C)；
     2. Peripheral blood leukocyte count ≥ 10000 /mm^3 or peripheral blood leukocyte count ≤ 4500 /mm^3 or peripheral blood rod-shaped granulocytes >15%.

Exclusion Criteria:

* Individuals who currently have epilepsy/myasthenia gravis or have a history of seizures (excluding febrile seizures in childhood)/myasthenia gravis history.
* Individuals undergoing hemodialysis or peritoneal dialysis.
* Invasive aspergillosis, mucormycosis, or other invasive fungal diseases.
* Current patients complicated with other infections, including endocarditis, osteomyelitis, central nervous system infection (such as meningitis, brain abscess, infection after cerebrospinal fluid shunt or shunt device infection), artificial joint infection, and active tuberculosis.
* It is currently complicated with refractory septic shock, and there was still persistent hypotension after sufficient fluid resuscitation or pressure therapy before randomization.
* Evidence of obvious liver disease or dysfunction, including known acute viral hepatitis or hepatic encephalopathy.
* Individuals with immunodeficiency or low immune function, including but not limited to: human immunodeficiency virus infection, hematological malignancies, bone marrow transplantation, immunosuppressive therapy, systemic corticosteroid therapy (defined as a daily dose equivalent to prednisone ≥ 20 mg and a course of treatment>14 days).
* Individuals with any laboratory test abnormalities during the screening period: aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) are 5 times higher than the upper limit of normal, or AST and/or ALT are 3 times higher than the upper limit of normal and total bilirubin is 1.5 times higher than the upper limit of normal, or neutrophil count is less than 1.0× 10^9/L or platelet count<60 ×10^9/L; Creatinine clearance rate ≤ 50 ml/min.
* According to the clinical judgment of the researchers, the expected survival period is less than 1 month.
* Individuals with allergic reactions to polymyxin or carbapenems.
* Subjects who require more than 2 systemic antibiotics for the treatment of Gram negative bacterial infections.
* Patients with acute physiology and chronic health (APACHE II) scores greater than 30.
* HAP/VAP subjects need to exclude:

  1. Patients with lung diseases that can interfere with treatment response evaluation, (such as cystic fibrosis, granulomatous diseases, pulmonary fungal infections, or recent pulmonary embolism);
  2. Individuals with lung abscess, empyema, or obstructive pneumonia;
  3. New York Heart Association (NYHA) Grade III-IV heart failure
  4. Lung or heart transplant recipients.
* CUTI subjects with/without pyelonephritis need to excluded:

  1. Subjects suspected or confirmed to have prostatitis;
  2. Renal transplant recipients;
  3. Individuals with ileal loops;
  4. Individuals who may continue to receive prophylactic treatment with antibiotics during clinical trials, such as those with bladder ureteral reflux;
  5. Patients that the indwelling catheter cannot be replaced during the study;
  6. Any unrecovered pelvic or urinary tract trauma;
  7. Individuals with simple urinary tract infections.
* cIAI subjects need to exclude:

  1. Upper gastrointestinal perforation, unless there is clear evidence of secondary infection in the abdominal cavity;
  2. Enrolled after surgery, but received over 1 dose of potentially effective systemic antibacterial medication before surgery.
* BSI subjects need to exclude:

  1. Subjects who only obtain positive blood culture through venous catheters (if both peripheral venous puncture blood culture and venous catheter blood culture show the same microbiological results, subjects can be selected);
  2. Infection is caused by intravascular sources, such as endocarditis, infected vascular grafts, and permanent intravascular devices that cannot be removed during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate (mITT) | At TOC visit, which is 7-14 days after the end of treatment.
  The proportion of patients in the modified intention to treat (mITT) population who achieved clinical cure at test of cure (TOC).

SECONDARY OUTCOMES:
Bacterial clearance rate | At TOC visit, which is 7-14 days after the end of treatment.
  Bacterial clearance rate of micro-MITT population at TOC visit
Clinical cure rate | At TOC visit, which is 7-14 days after the end of treatment.
  The proportion of subjects with clinical evaluation of clinical cure at the TOC visit. Clinical cure refers to the following: The symptoms, signs, and laboratory test abnormalities of the subjects who were infected after the end of treatment have all returned to normal or pre-infection status, and no new symptoms, signs, or laboratory test abnormalities have occurred, nor have complications occurred.
Microbiological efficacy | At TOC visit, which is 7-14 days after the end of treatment.
  The proportion of subjects with effective microbial efficacy evaluation (microbial clearance or presumed clearance, including bacterial population alternation, which is also classified as clearance) according to subject evaluation and pathogen evaluation during the TOC visit.
All-cause mortality rate | 28±2 days after randomization.
  The all-cause mortality rate at 28±2 days in the mITT population
Peak concentration (Cmax) | 72 hours before the first dose; 30 minutes before the first dose, at the end and 2, 4, 6, 8 hours after dose on day 4; 30 minutes before the second dose; 30 minutes before the first dose on day 10.
  Maximum plasma drug concentration
Peak time (Tmax) | 72 hours before the first dose; 30 minutes before the first dose, at the end and 2, 4, 6, 8 hours after dose on day 4; 30 minutes before the second dose; 30 minutes before the first dose on day 10.
  Time to reach maximum plasma drug concentration

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The People's Hospital of Chizhou, Chizhou, Anhui
  - Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - People's Hospital of Chongqing Banan District, Chongqing, Chongqing Municipality
  - Chongqing University Jiangjin Hospital, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University School of Medicine, Shantou, Guangdong
  - Luoyang Central Hospital, Luoyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Changsha Central Hospital, Changsha, Hunan
  - Huai'an Second People's Hospital, Huaian, Jiangsu
  - General Hospital of the Eastern Theater Command, Nanjing, Jiangsu
  - Taizhou Hospital of TCM, Taizhou, Jiangsu
  - Jiangsu Subei People's Hospital, Yangzhou, Jiangsu
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huadong Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiading District Central Hospital, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang